CLINICAL TRIAL: NCT05303883
Title: Feasibility of Pediatric Constraint Induced Movement Therapy Delivered Remotely for Children With Hemiplegic Cerebral Palsy
Brief Title: Feasibility of Pediatric CIMT by Televideo
Acronym: CHAMP-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Amy Darragh, Director of the Occupational Therapy Division in the School of Health and Rehabilitation Sciences in the College of Medicine, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001867
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Motor impairments; Gross motor delays; Manual impairment; Upper extremity impairment

STUDY DESIGN:
Intervention Model Description: All enrolled children will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric constraint induced therapy (Experimental): Constrained induced therapy for children with hemiplegic cerebral palsy. Three hours of therapy per day, for five days a week, for four weeks.
  Interventions: Other: Pediatric Constrained Induced Movement Therapy

INTERVENTIONS:
Other: Pediatric Constrained Induced Movement Therapy — Constraint of the child's less-impaired upper extremity for first 17 days of treatment. Children wear a removable, lightweight constraint for the first 17 of 20 therapy sessions.

SUMMARY:
The study will test a remotely delivered, intensive, therapist-led, pediatric CIMT intervention, to improve the quality and frequency of upper limb movement during functional activity. We will evaluate: remote assessment of patient motor outcomes; computer-based video interaction for parent training in shaping therapeutic activities; child, parent, and therapist interactions; remote delivery of treatment; and the usability and usefulness of technology (e.g. reliability of internet connection; video streaming). As a final product, the study will yield a feasible and acceptable tele-rehabilitation protocol that meets our fidelity and reliability criteria and is ready for larger-scale efficacy testing in children with hemiplegic CP, ages 1-10 years.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a public health problem that affects 2-3 per 1000 children. Up to 75 % of children with cerebral palsy will have motor impairments that can lead to lifelong disability, therefore there is a need for effective treatment of these motor impairments. A body of evidence shows that intensive motor therapies can improve arm and hand (upper limb) motor function in children with CP. Constraint induced movement therapy (CIMT) is one of the motor therapies with the strongest evidence base for its effectiveness. Our team has developed an innovative CIMT protocol to treat upper limb impairments due to CP. This protocol combines 1) high dosage of motor treatments, (up to 3-6 hours of therapy per day for 20 days); 2) constraint of the unaffected arm, 3) the incorporation of behavior motivation techniques to encourage the child to perform increasingly complex motor tasks; 4) treatment within the home to promote generalization of the motor behaviors; and 5) a post-therapy treatment plan for the parents to continue after the formal CIMT protocol is done. In a recent randomized controlled trial, we tested the effect of this CIMT protocol on upper limb function in children with hemiplegic CP. Children who received CIMT at the 30-hour and 60-hour doses had significantly better function immediately post-treatment than children who received usual and customary care. This difference persisted at 6 months after treatment for the children who received the 60-hour dose. These results provide clear evidence that the higher therapy dose resulted in greater sustained improvement of upper limb function.

Through our work in this and other clinical trials, we recognized that our treatment protocol delivered in the home cannot be delivered to children who live in rural areas beyond the reach of our therapists or in urban communities whose families are unable to have therapists work in their homes for 20 days. This limitation disproportionately affects families who live in medically resource poor areas. To address this barrier to access, we propose to modify our CIMT protocol so it can be used for telehealth delivery. Rehabilitation by telehealth has drawn considerable attention in the adult stroke world. A small number of trials in adult stroke patients and a small pilot trial in pediatric patients with upper limb weakness have shown that upper limb rehabilitation by telehealth is feasible and can be as effective as that delivered in the clinic.

Based on this emerging evidence, we will test the feasibility of our CIMT protocol adapted for telerehabilitation. In a related study, we will refine our CIMT by soliciting the input of families and children who have undergone CIMT treatment, and the input of expert treating therapists and assessors regarding our protocol. In the current study, we will test this refined protocol in a pilot sample of five to seven children ages 1-10 years who have hemiplegic CP. We will evaluate whether the remotely delivered treatment maintains fidelity to the original version delivered in person; whether the treatment is feasible to deliver, and whether it is acceptable to families, therapists, and assessors. In addition, we will evaluate whether the remote assessment of fine and gross motor skills is feasible, reliable, and acceptable. These measures will be assessed by questionnaires, observation of assessment recordings, scoring of the outcome measure, and interviews of parents of and participating children (the primary stakeholders), as well as feedback from study assessors.

Our long-term goal is to implement effective, accessible, intensive upper-limb interventions for children with hemiparesis, using delivery methods that are accessible, available, and feasible for families representing socioeconomic, geographic, and racial/ethnic diversity. This clinical research study is an important step toward clinical implementation through translation of an evidence-based intervention to a potentially more accessible, practical and equitable delivery method for families of children with CP.

ELIGIBILITY:
Inclusion Criteria:

1. ages 1 - 10 years old at enrollment;
2. diagnosis of hemiplegic CP per parent report;
3. ability to participate in therapy 3 hours/day x 5 days/week x 4 weeks (dose based on CHAMP RCT results).

Exclusion Criteria:

1. uncontrolled seizures;
2. medical or other complex conditions that preclude tolerance of 3 hours of intensive therapy per day

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Within 2 weeks of intervention completion
  The Feasibility of Intervention Measure (FIM) will assess intervention feasibility with a four-item measure. The measure includes four statements about the plausibility of implementing the intervention (the intervention seems implementable; the intervention seems doable; the intervention seems possible; the intervention seems easy to use). Individuals rate the extent to which the agree with each statement on a five-level scale (completely disagree, disagree, neither agree or disagree, agree, completely agree).
Acceptability of Intervention Measure (AIM) | Within 2 weeks of intervention completion
  Acceptability of Intervention will be assessed through a four-item measure (AIM). The measure includes four statements about the appeal of the intervention (e.g. I like the intervention; I welcome the intervention; the intervention meets my approval; the intervention is appealing to me). Individuals rate the extent to which the agree with each statement on a five-level scale (completely disagree, disagree, neither agree or disagree, agree, completely agree).
Intervention Appropriateness Measure (IAM) | Within 2 weeks of intervention completion
  Intervention Appropriateness will be assessed through a four-item measure (IAM). The measure includes four statements about the relevance or pertinence of the intervention (e.g. the intervention seems suitable; the intervention seems applicable; the intervention seems fitting; the intervention seems like a good match). Individuals rate the extent to which the agree with each statement on a five-level scale (completely disagree, disagree, neither agree or disagree, agree, completely agree).
Usefulness, Usability and Desirability Assessment (UUD) | Within 2 weeks of intervention completion
  The Usability of the remote delivery system (use of the iPad, Kubi robot; video upload) will be assessed with the UUD assessment. Usability includes three major components: usefulness, desirability, and usability. The UUD gathers data on usability (ease of use of the telehealth technology) (9 items), usefulness (value, relevance, and applicability of the telehealth technology) (10 items), and desirability (overall appeal or interest of the telehealth technology) (4 items). Items are rated a five-point Likert-type scale.
Fidelity of Intervention Assessment | Once per week during 4-week intervention period
  This instrument assesses the extent to which the therapist adhered to fifteen core constructs of the intervention protocol. Evidence of adherence to high quality pediatric rehabilitation elements includes 6 constructs that are scored as Present (present-some and present-strong) or Absent. Includes items such as "collaboration between parent and therapist" and "aligning therapy with child's goals". Evidence of core components of pediatric constraint induced movement therapy is scored as Present or Absent. Includes items such as "high intensity of intervention" and occurs in "natural environment". Total score is number of core components present.

SECONDARY OUTCOMES:
Fidelity of Remote Assessment | Within one week following the assessment
  Fidelity to remote assessment procedures will be determined through video coding of recorded remote assessment. The following will be coded: adherence to administration procedures, length of assessment, number of sessions to complete assessment, number of assessment items completed, and percentage of items completed.
Perceptions of Remote Assessment and Intervention | Within one week following the intervention.
  A semi-structured interview will be used to assess the perceptions of therapists, assessors, and parents about the process of remote delivery. There are fourteen open-ended questions about the remote assessment process, the remote intervention process, and the technology used to gather information and conduct the remote assessments and intervention. These will will be coded qualitatively and analyzed by content analysis to determine common perceptions of strengths and areas for improvement.

OTHER OUTCOMES:
Parent therapist information exchange | Within 1 week following intervention
  This measures assesses the satisfaction regarding communication between the therapist and the family, with particular emphasis on preparation of the parent for engaging with their child during therapy activities.. The measures includes 21 questions rated on a four-point scale about the parent role in therapy, the preparation and training for parent participation in therapy, and goal setting. Additional questions ask for a description of the characteristics that the parent role, what were positive experiences with the parent-therapist relationship, and suggestions for how to improve the therapist-parent relationship.
Abilhand-kids | Within 2 weeks prior to start of intervention and within 1 week following intervention
  ABILHAND-kids is a parent reported measure of manual ability in children with Cerebral Palsy. Parents estimate their child's ease/difficulty with performing 21 selected activities of daily living. Parents rate their child's difficulty on a three-level scale: "Impossible", "Difficult", or "Easy".
Box and Block | Within 2 weeks prior to start of intervention and within 1 week following intervention
  The Box and Block assesses manual dexterity. It has strong psychometric properties. The child is instructed to move 1-inch square blocks from one side of a wooden box over a partition to the other side. The scoring is based on the number of blocks moved over within 60 seconds.
Structured Activity Session | Within 2 weeks prior to start of intervention and within 1 week following intervention
  The Structured Activity Session identifies a variety of age-appropriate activities and behaviors that can be coded for quality and frequency of movement, as well as the number of activities and behaviors completed. The activity session will include a 1. dressing activity (e.g. donning and doffing and zippered sweatshirt), 2. a snack activity (e.g. opening a beverage container, opening and eating a snack with small food items like goldfish, and opening and eating a snack with a utensil like applesauce or pudding), and gross motor activities (like catching a ball, jumping).

CONTACTS AND LOCATIONS:
Overall Officials: Warren Lo, Principal Investigator — Nationwide Children's Hospital; Amy Darragh, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Virginia Polytechnic Institute and State University, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No